CLINICAL TRIAL: NCT00456131
Title: Prevention of Obesity at Universities: A Randomized Trial
Acronym: Healthy Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Lowe, Principal Investigator, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK72982; R01DK072982 (NIH)
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): The intervention group (other group is a control without any intervention) involves 6 one-hour group sessions teaching healthy eating habits and weight gain prevention tools.
  Interventions: Behavioral: Healthy Eating Behaviors Training

INTERVENTIONS:
Behavioral: Healthy Eating Behaviors Training — The intervention group (other group is a control without any intervention) involves 6 one-hour group sessions teaching healthy eating habits and weight gain prevention tools.

SUMMARY:
This is a nutrition and behavior-based intervention conducted at Drexel University and the University of Pennsylvania with college women during their freshman year. It involves attending groups where life skills and eating behaviors are taught to help them control their weight and physical health.

ELIGIBILITY:
Inclusion Criteria:

* A variety of risk factors for later life weight gain

Exclusion Criteria:

* Current or past history of eating disorder

Ages: 18 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2006-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Weight | baseline, 6 weeks, 6 months, 12 months, 24 months
blood work | baseline, 6 months, 24 months
questionnaire data | baseline, 6 weeks, 6 months, 12 months, 24 months
Body Composition | baseline, 6 months, 24 months

SECONDARY OUTCOMES:
dietary recalls | baseline, 6 weeks, 6 months, 12 months, 24 months
Pedometer readings | baseline, 6 weeks, 6 months, 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Low, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Phildadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Lowe MR, Feig EH, Winter SR, Stice E. Short-term variability in body weight predicts long-term weight gain. Am J Clin Nutr. 2015 Nov;102(5):995-9. doi: 10.3945/ajcn.115.115402. Epub 2015 Sep 9. PMID 26354535
- [Derived] Berner LA, Arigo D, Mayer LE, Sarwer DB, Lowe MR. Examination of central body fat deposition as a risk factor for loss-of-control eating. Am J Clin Nutr. 2015 Oct;102(4):736-44. doi: 10.3945/ajcn.115.107128. Epub 2015 Sep 9. PMID 26354534